CLINICAL TRIAL: NCT04890379
Title: Dimethyl Fumarate for the Treatment of Intracerebral Hemorrhage
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: There are no sufficient patients in the hospital.
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: haojunwei2
Record Dates: First submitted 2021-05-10; First posted 2021-05-18 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2021-05

CONDITIONS: Intracerebral Hemorrhage
Keywords: Dimethyl Fumarate; Intracerebral Hemorrhage(ICH); perihematomal edema(PHE); neurologic deficit; immune modulator
MeSH Terms: conditions — Cerebral Hemorrhage; Neurologic Manifestations | interventions — Dimethyl Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard management plus Dimethyl Fumarate (Experimental)
  Interventions: Drug: Dimethyl fumarate
- standard management plus placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dimethyl fumarate — Dimethyl fumarate 240mg orally twice daily for 3 consecutive days
  Arms: standard management plus Dimethyl Fumarate
Drug: Placebo — Placebo 240mg orally twice daily for 3 consecutive days
  Arms: standard management plus placebo

SUMMARY:
The investigators conduct this study to investigate whether oral administration of Dimethyl Fumarate, a Food and Drug Administration-approved drug for multiple sclerosis, is safe and effective in alleviating PHE and neurologic deficits in patients with ICH.

ELIGIBILITY:
Inclusion Criteria:

1. Men and nonpregnant women aged 18 years and older
2. a primary supratentorial ICH of 5 to 30 mL
3. symptom onset less than 72 hours prior to admission
4. a Glasgow Coma Scale (GCS) score of 6 or greater
5. basal ganglia hemorrhage only

Exclusion Criteria:

1. patients with a GCS score of 3 to 5
2. planned surgical evacuation of a large hematoma (>30 mL)
3. various degrees of dysphagia,and nausea/vomiting, any of which renders oral administration of fingolimod difficult
4. patients with hematoma expansion
5. secondary ICH
6. preexisting disability (modified Rankin Scale [mRS] score >1)
7. any history of bradycardia or atrioventricular block
8. concomitant use of antineoplastic, immunosuppressive, or immune-modulating therapies
9. macular edema
10. Patients with known hypersensitivity to dimethyl fumarate or to any excipient of this product
11. Pregnant and lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Volume of Perihematomal edema(PHE) | day7
  measured by MRI
Glasgow Coma Scale (GCS) | day7
  The GCS score ranges from 3 to 15 points. The lower the score, the more severe the patient's coma is.
National Institutes of Health Stroke Scale (NIHSS) | day 7
  The NIHSS score ranges from 0 to 42 points. The higher the score, the more severe the neurological impairment.

SECONDARY OUTCOMES:
Volume of Perihematomal edema(PHE) | day1
  measured by MRI
Volume of Perihematomal edema(PHE) | day3
  measured by MRI
Volume of Perihematomal edema(PHE) | day14
  measured by MRI
Volume of Perihematomal edema(PHE) | day90
  measured by MRI
Glasgow Coma Scale (GCS) | day 1
  The GCS score ranges from 3 to 15 points. The lower the score, the more severe the patient's coma is.
Glasgow Coma Scale (GCS) | day 3
  The GCS score ranges from 3 to 15 points. The lower the score, the more severe the patient's coma is.
Glasgow Coma Scale (GCS) | day 14
  The GCS score ranges from 3 to 15 points. The lower the score, the more severe the patient's coma is.
National Institutes of Health Stroke Scale (NIHSS) | day1
  The NIHSS score ranges from 0 to 42 points. The higher the score, the more severe the neurological impairment.
National Institutes of Health Stroke Scale (NIHSS) | day3
  The NIHSS score ranges from 0 to 42 points. The higher the score, the more severe the neurological impairment.
National Institutes of Health Stroke Scale (NIHSS) | day14
  The NIHSS score ranges from 0 to 42 points. The higher the score, the more severe the neurological impairment.
National Institutes of Health Stroke Scale (NIHSS) | day90
  The NIHSS score ranges from 0 to 42 points. The higher the score, the more severe the neurological impairment.
The Modified Rankin Scale (mRS) | day1
  The mRS score ranges from 0 to 7 points. The higher the score, the more severe the neurological recovery state of stroke patients.
The Modified Rankin Scale (mRS) | day3
  The mRS score ranges from 0 to 7 points. The higher the score, the more severe the neurological recovery state of stroke patients.
The Modified Rankin Scale (mRS) | day7
  The mRS score ranges from 0 to 7 points. The higher the score, the more severe the neurological recovery state of stroke patients.
The Modified Rankin Scale (mRS) | day14
  The mRS score ranges from 0 to 7 points. The higher the score, the more severe the neurological recovery state of stroke patients.
The Modified Rankin Scale (mRS) | day90
  The mRS score ranges from 0 to 7 points. The higher the score, the more severe the neurological recovery state of stroke patients.
The Modified Barthel Index (mBI) | day 1
  The mBI score ranges from 0 to 100 points. The higher the score, the higher the degree of independence of stroke patients.
The Modified Barthel Index (mBI) | day 3
  The mBI score ranges from 0 to 100 points. The higher the score, the higher the degree of independence of stroke patients.
The Modified Barthel Index (mBI) | day 7
  The mBI score ranges from 0 to 100 points. The higher the score, the higher the degree of independence of stroke patients.
The Modified Barthel Index (mBI) | day 14
  The mBI score ranges from 0 to 100 points. The higher the score, the higher the degree of independence of stroke patients.
The Modified Barthel Index (mBI) | day 90
  The mBI score ranges from 0 to 100 points. The higher the score, the higher the degree of independence of stroke patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Beijing, Beijing, Beijing Municipality, China